CLINICAL TRIAL: NCT05647551
Title: A Prospective, Open-Label Study to Evaluate Subject's Satisfaction With the Aesthetics of the Periorbital Area After Treatment of the Upper and/or Mid Face With JUVÉDERM® Fillers and BOTOX®/VISTABEL®
Brief Title: A Study to Evaluate Satisfaction in Adult Participants With the Aesthetics of the Periorbital Area After JUVÉDERM® Fillers and BOTOX®/VISTABEL® Injections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M22-979; 2022-000417-13 (EudraCT Number)
Record Dates: First submitted 2022-12-09; First posted 2022-12-12 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Facial Corrections; Facial Lines
Keywords: JUVÉDERM fillers; BOTOX/VISTABEL

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- JUVÉDERM fillers and BOTOX/VISTABEL (Experimental): At Visit 1, JUVÉDERM filler injections (Juvéderm VOLBELLA with lidocaine, Juvéderm VOLIFT with lidocaine, and/or Juvéderm VOLUMA with lidocaine) will be administered. At Visit 4, JUVÉDERM VOLBELLA with lidocaine, may be administered in the infraorbital hollow (IOH)/tear trough (TT) area. At Visit 6, participants will receive BOTOX/VISTABEL. Touch-ups may be performed as required based on investigator's assessment.
  Interventions: Drug: BOTOX®/VISTABEL®; Device: Juvéderm® VOLBELLA® with Lidocaine; Device: Juvéderm® VOLIFT® with Lidocaine; Device: Juvéderm® VOLUMA® with Lidocaine

INTERVENTIONS:
Drug: BOTOX®/VISTABEL® — Facial Injection
Device: Juvéderm® VOLBELLA® with Lidocaine — Facial Injection
Device: Juvéderm® VOLIFT® with Lidocaine — Facial Injection
Device: Juvéderm® VOLUMA® with Lidocaine — Facial Injection

SUMMARY:
Different studies have shown the negative effects of aging around the area of the eyes. Signs of aging may contribute to erroneously projected emotions (e.g., anger, tiredness, or sadness) that do not reflect the individual's true feelings affecting interpersonal relationships. Minimally invasive aesthetic treatments with botulinum toxin and hyaluronic acid (HA) fillers are used to treat wrinkles and volume deficiencies associated with the appearance of most of the signs of aging.

This Phase 4 post-marketing study is an open-label study in which all subjects will receive active study treatment. The purpose of this study is to evaluate the subject's satisfaction after the treatment of JUVÉDERM® fillers and BOTOX®/VISTABEL® on the upper and/or mid face, which includes areas around the eyes, under the eyes, eyebrows, the temple, and the cheek.

This study will enroll approximately 80 healthy male and female subjects ages 40 to 65 across 10 sites in Australia, Belgium, and United Kingdom. Each subject will be in the study for approximately 90 days. The initial treatment of the JUVÉDERM fillers (Juvéderm VOLBELLA with lidocaine, Juvéderm VOLIFT with lidocaine, and/ or Juvéderm VOLUMA with lidocaine) will be given on Visit 2, and if needed, a touch-up treatment will be given. On Visit 4, the Juvéderm VOLBELLA with lidocaine filler, may be given, followed by a touch-up treatment, if needed. On Visit 6, subjects will receive study drug BOTOX/VISTABEL. All subjects will return for the study exit visit on Day 90.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, checking for side effects, and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participant's dissatisfaction with eyes, measured by a baseline score of "very dissatisfied" or "somewhat dissatisfied" in at least 3 of the 7 items in the FACE-Q Satisfaction with Eyes.
* Have some degree of IOH/TT per Allergan Infraorbital Hollows Scale (AIHS) (1 [minimal], 2 [moderate], 3 [severe], or 4 [extreme]) on both sides with a chance of improvement either by direct or indirect treatment, per investigator's assessment.
* Need for treatment in at least 2 areas in the upper and/or mid face (e.g., eyebrows, IOH/TT, temples, malar or zygomatic, fine lines such as periorbital lines), with at least two of the JUVÉDERM products (Juvéderm VOLBELLA, Juvéderm VOLIFT, or Juvéderm VOLUMA), per investigator's assessment.
* Participant meets at least one of the following criteria (investigator's assessment):

  * 2 or 3 (moderate or severe) on Allergan Glabellar Lines Severity Scale at maximum furrow.
  * 2 or 3 (moderate or severe) on Lateral Canthal Lines Severity Scale at maximum smile.
* Participants must have a score of ≥ 5 for Facial Line Outcomes-11 item 1 (Bothered by Facial Lines).

Exclusion Criteria:

* Participants with presence of inflammation, infection at any injection site or systemic infection (study entry may be postponed until one week following recovery), noticeable acne scarring, cancerous or pre-cancerous lesion, or unhealed wound or have undergone radiation treatment in the area to be treated.
* Participant with an allergy or sensitivity to investigational products or their components.
* Participant with history or current symptoms of dysphagia.
* Participant has medical condition that may increase the risk of exposure to botulinum toxin including diagnosed myasthenia gravis, Eaton-Lambert Syndrome, amyotrophic lateral sclerosis, or any other disease that might interfere with neuromuscular function.
* Participant has profound atrophy/excessive weakness of muscles in target areas of injection.
* Participant has marked facial asymmetry, brow or eyelid ptosis, excessive dermatochalasis, deep dermal scarring, thick sebaceous skin, or an inability to substantially lessen the resting Glabellar Lines (GLs) and Lateral Canthal Lines (LCLs)/facial rhytides by physically spreading them apart.
* Participant has tendency to accumulate fluid in the lower eyelids, or large infraorbital fat pads, i.e., significant convexity or projection from the infraorbital fat pads that would mask improvement.
* Participant has mid face volume deficit due to congenital defect, trauma, abnormalities in adipose tissue related to immune-mediated diseases such as generalized lipodystrophy (e.g., juvenile dermatomyositis), partial lipodystrophy (e.g., Barraquer-Simons syndrome), inherited disease, or human immunodeficiency virus-related disease.
* Participant has undergone live vaccination, surgery, or dental procedures (e.g., tooth extraction, orthodontia, or implantation) within 30 days prior to enrollment or be planning to undergo any of these procedures during the study and up to 30 days after the study.
* Participant has neuromuscular disorders including generalized muscle weakness, diplopia, ptosis, dysphonia, dysarthria, severe dysphagia, and respiratory compromise.
* Participant has received temporary or semi-permanent filler injections at upper or mid face (e.g., HA, calcium hydroxyapatite, L-polylactic acid) within 2 years prior to entry in the study.
* Participant has received any investigational product or device within 30 days or 5 half-lives of the drug (whichever is longer) prior to study enrollment or planning to participate in another investigation during the course of this study.
* Participant has undergone at anytime plastic surgery of the face, tissue grafting, or tissue augmentation with silicone, fat, or other permanent dermal fillers, or be planning to undergo any of these procedures at any time during the study.
* Participant has received mesotherapy, skin resurfacing (laser, photomodulation, intense pulsed light, radio frequency, dermabrasion, chemical peel, or non-ablative procedures) in the face within 6 months prior to study enrollment.
* Participant has a current use of nonsteroidal anti-inflammatory drug (e.g., aspirin, ibuprofen) with the exception of a daily low dose of aspirin, from 10 days prior to injection up to 3 days post-injection.
* Participant has had topical retinoid therapy and/or topical hormone cream applied to the face, for potential participants who have not been on a consistent dose regimen for at least 6 months prior to enrollment and who are unable to maintain regimen for the study.
* Participant has received systemic retinoid therapy within one year prior to study enrollment.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the overall score of the participant's FACE-Q™ Satisfaction with Eyes with JUVÉDERM fillers and BOTOX/VISTABEL | Up to 90 Days
  The FACE-Q Satisfaction with Eyes is a 7-item scale with a 4-point response options ranging from "very dissatisfied" to "very satisfied". The responses will be summed and converted to a Rasch transformed score that ranges from 0 to 100. Higher scores indicate higher satisfaction.

SECONDARY OUTCOMES:
Percentage of Participants Achieving "Responder" status based on participant's assessment of GAIS of periorbital area | At Day 90
  The GAIS uses a 5-point scale where: 2=much improved, 1=improved, 0=no change, -1=worse and -2=much worse. A responder is defined as "improved" or "much improved" in the overall aesthetics assessment in the periorbital area.
Percentage of Participant Achieving "Responder" status based on investigator's assessment of GAIS of periorbital area | at Day 90
  The GAIS uses a 5-point scale where: 2=much improved, 1=improved, 0=no change, -1=worse and -2=much worse. A responder is defined as "improved" or "much improved" in the overall aesthetics assessment in the periorbital area.
Percentage of Participants Achieving "Responder" status based on investigator's assessment of global aesthetic improvement scale (GAIS) of infraorbital area | At Day 30
  The GAIS uses a 5-point scale where: 2=much improved, 1=improved, 0=no change, -1=worse and -2=much worse. A responder is defined as "improved" or "much improved" in the overall aesthetics assessment in the infraorbital area.
Change from baseline in overall score of the participant's assessment of FACE-Q Psychological Function | Up to 90 Days
  The FACE-Q Psychological Function is a 10-item scale that measures psychological function with a 4-point response options ranging from "definitely disagree" to "definitely agree". The responses will be summed and converted to a Rasch transformed score that ranges from 0 to 100. Higher scores indicate higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (8):
- Australia (4):
  - Eastern Plastic Surgery /ID# 244785, Box Hill North, Victoria
  - Dermatology Institute of Victoria /ID# 244786, South Yarra, Victoria
  - Complete Skin Specialists /ID# 244840, Sunbury, Victoria
  - SkinBox Clinics /ID# 244787, Fremantle
- Belgium (4):
  - UZ Brussel /ID# 244761, Jette, Brussels Capital
  - Centre de la fontaine /ID# 244763, Gerpinnes, Hainaut
  - Plastische Chirurgie B V /ID# 253395, Oudenaarde, Oost-Vlaanderen
  - Duinbergen Clinic /ID# 244765, Knokke-Heist, West-Vlaanderen

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=M22-979#additional-resources-section